CLINICAL TRIAL: NCT05264532
Title: BRCAShare: Video Intervention for Relatives of BRCA Mutation-Positive Patients
Brief Title: Usefulness of Video-Based Intervention in Helping Participants Encourage Their Families to Get Tested for BRCA Gene Mutations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Leigha Senter-Jamieson, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-17312; NCI-2018-00756 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-06-25; First posted 2022-03-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: BRCA1 Gene Mutation; BRCA2 Gene Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (video via text message) (Experimental): Participants receive a 2-minute information-graphic video via text message consisting of misconceptions and issues that may be paramount when discussing mutation status with relatives that they can share with family via text message, email, or social media.
  Interventions: Other: Informational Intervention; Other: Survey Administration
- Arm B (letter via standard U.S. mail) (Active Comparator): Participants receive family letter via U.S. postal service mail consisting of misconceptions and issues that may be paramount when discussing mutation status with relatives.
  Interventions: Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Receive information-graphic video
  Arms: Arm A (video via text message)
Other: Informational Intervention — Receive family letter
  Arms: Arm B (letter via standard U.S. mail)
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies how well a video-based intervention works in helping participants encourage their families to get tested for BRCA gene mutations. Testing in families with BRCA gene mutations can allow for risk management and reduction with the overall goal of reducing cancer burden. Video-based intervention sent via text messages may help participants easily share information about BRCA gene mutations with family members.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To understand whether the use of a video-based message to encourage cascade testing, delivered via short message service (SMS) (text message) or shared on social media, is superior to a written message as a method of information-sharing among families that have BRCA gene mutations.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Participants receive a 2-minute information-graphic video via text message consisting of misconceptions and issues that may be paramount when discussing mutation status with relatives that they can share with family via text message, email, or social media.

ARM B: Participants receive family letter via U.S. postal service mail consisting of misconceptions and issues that may be paramount when discussing mutation status with relatives.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who test positive for mutations in BRCA1 or BRCA2 are eligible for this study
* Family members who receive the video message/family letter will be invited to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Impact of a web-based video delivered via text message or shared on social media on information sharing among relatives belonging to families with BRCA gene mutations | Up to 3 years
  Measure participant-reported information sharing among family members prior to receipt of the video and after the video. There is no previously validated scale/set of items for this. Items are investigator created and assess likelihood to share information with family members on a Likert scale.
Impact of participant-reported family dynamics on information sharing | Up to 3 years
  Brief family relationship scale will be used to determine whether differences in family dynamics could be associated with differences in family sharing. A higher score for the cohesion and expressiveness subscales generally indicates more positive dynamics and a the conflict subscale is inversely scored.

CONTACTS AND LOCATIONS:
Overall Officials: Leigha Senter, LGC, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu